CLINICAL TRIAL: NCT06098846
Title: Double-Blind Placebo-Controlled Human Transdermal Vitamin D Supplement Study
Brief Title: Human Transdermal Vitamin D Supplement Study
Acronym: TransVitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Vitamax Wholesalers LLP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR/DP-22/23-34078
Record Dates: First submitted 2023-10-05; First posted 2023-10-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Supplementation
Keywords: vitamin D; supplementation; transdermal patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo patch (Placebo Comparator): Placebo transdermal patch daily
  Interventions: Dietary Supplement: Placebo transdermal patch
- Dose Frequency 1 (Active Comparator): Active transdermal patch daily (actives could be alternated with placebo in a given sequence)
  Interventions: Dietary Supplement: Vitamin D phosphate
- Dose Frequency 2 (Active Comparator): Active transdermal patch daily (actives could be alternated with placebo in a given sequence)
  Interventions: Dietary Supplement: Vitamin D phosphate
- Dose Frequency 3 (Active Comparator): Active transdermal patch daily (actives could be alternated with placebo in a given sequence)
  Interventions: Dietary Supplement: Vitamin D phosphate

INTERVENTIONS:
Dietary Supplement: Vitamin D phosphate — Application of a Vitamin D phosphate active patch
  Arms: Dose Frequency 1; Dose Frequency 2; Dose Frequency 3
Dietary Supplement: Placebo transdermal patch — Application of a placebo transdermal patch
  Arms: Placebo patch

SUMMARY:
Despite the wide availability of vitamin D supplements vitamin D deficiency remains a concerning global problem. It is hypothesised that hypothesize that vitamin D delivered via the skin will overcome the problems associated with variable oral bioavailability and lead to a patient-friendly and efficacious means to supplement this vitamin. The main objective of this study is therefore to test the efficacy of a vitamin D transdermal patch that employs vitamin D phosphate to deliver the vitamin D into the blood.

In this two-part supplementation study healthy individuals with a risk of vitamin D deficiency (n=118), aged between 18 - 65 years, will be recruited. The recruitment in central London, UK, will ensure a multicultural, multi-ethnic cohort to enable the findings to be translated into evidence to try and find a solution for the global vitamin D deficiency problem.

DETAILED DESCRIPTION:
The primary objective of this study is to understand the ability of a vitamin D transdermal patch to provide effective vitamin D supplementation. To do this, the study team will identify, using a questionnaire (validated collection tool), a cohort of healthy individuals who are at risk of vitamin D deficiency. The study team will take the personal details of the volunteers, a full medical history, food, exercise, body indices, and diet information and register these details. A baseline assessment will be taken of those patients who are identified by the questionnaire as likely to have low vitamin D levels and meet the study inclusion and exclusion criteria. The baseline measurements will include a blood sample to determine 25(OH)vitamin D3 (25(OH)VD3) concentration in the serum (perhaps also other metabolites), vitamin D binding protein (VDBP) concentrations in the blood serum and the skin interstitial fluid, parathyroid hormone levels and calcium in the blood. It will also require images of the human nails. This information will help to understand the vitamin D status of each study participant. This baseline data will be uploaded to a secure database and form the basic demographic information and baseline levels prior to the application of the vitamin D supplement patch.

The supplementation study will take 2 parts. In part one, two cohorts of 8 participants will be provided with one of two doses of the supplement in a dose escalation pilot study. These cohorts will be supplemented in sequence to establish the safety of the dose, with the lowest dose being confirmed to be safe prior to the second dose being tested. The primary outcome will be safety and tolerability. A calcium measure of more than 12 mg/dL or 25(OH)VD3 > 150 nM/L will indicate a risk of toxicity at the 2-week or 4-week blood draw and the dosing would terminate and this would be considered as a serious adverse event. If there are serious adverse events in 2 or more of the participants the dose will not be safe. The secondary outcome will be efficacy, and a change of 25(OH)VD3 of less than 5 nM/L in more than 75% of participants would indicate the dose is ineffective after 4 weeks and this will be used to guide the second cohort dosing.

Upon completion of part 1 the second part will begin. In part 2, the participants will be randomized by a statistician into 4 interventional arms, one placebo, and 3 different patch dosing frequencies. In part 2, the study will last 8 weeks with measurements at weeks 4 and 8. Part 2 will have an interim analysis at week 4, then it will proceed with only 2 study arms and make final measurements on week 8. The dosing for part 2 in the different arms of the study will be based on the part 1 results. The aim of these two studies is to establish if vitamin D supplementation via the skin improves the vitamin D status and at what dosing level/interval is required to achieve this.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 18 and 65 years of age
2. Suspected low vitamin D levels (defined as moderate or high risk using the Deschasaux questionnaire (10))
3. Written informed consent for study participation.
4. Willingness to comply with all study requirements.
5. Competent use of English language.

Exclusion Criteria:

1. Patients unable to give informed consent.
2. The use of vitamin D supplements 4 weeks prior to the commencement of the study (and unwilling to washout).
3. Pregnancy
4. Those with parathyroid, thyroid, or calcium disorders, sarcoidosis, a requirement for calcium channel blockers, Type I diabetes, and concurrent active malignancies.
5. Those who have been diagnosed with vitamin D deficiency by a GP in the last 3 months using a blood test.
6. Those who have been diagnosed with vitamin D deficiency by a GP in the last 6 months using a blood test and have not taken any vitamin D supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the % change in 25(OH)vitamin D3 concentration in human serum compared to baseline | After 4 and 8 weeks compared to baseline
  Concentration of 25(OH)vitamin in the serum (ng/ml)

SECONDARY OUTCOMES:
Measurement of the % change in vitamin D binding protein concentration in human serum compared to baseline | After 4 and 8 weeks compared to baseline
  Concentration of vitamin D binding protein levels in the serum (micrograms per ml)
Measurement % of chemical biomarker concentrations in the human skin interstitial fluid compared to baseline | 4 and 8 weeks compared to baseline
  Concentration change of chemicals identified in skin interstitial fluid (ng/ml)
Measurement of the change in human nail plate characteristics measured using pixels compared to baseline | 4 and 8 weeks compared to baseline
  Quantification of image feature change in nail photographs (unit pixels)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Jones, Principal Investigator — King's College London
Locations (1):
- Institute of Pharmaceutical Science, King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hibbard T, Andriollo P, Lim CH, Guo Q, Lawrence KP, Coker B, Malek R, Douiri A, Alhnan MA, Jones SA. A multistage double-blind placebo-controlled study to assess the safety and efficacy of transdermal vitamin D phosphate supplementation (TransVitD). Trials. 2025 Feb 19;26(1):59. doi: 10.1186/s13063-024-08711-8. PMID 39972355